CLINICAL TRIAL: NCT00671294
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Determine the Safety and Efficacy of TAK-375 in Elderly Subjects With Chronic Insomnia.
Brief Title: Safety and Efficacy of Ramelteon in Elderly Subjects With Chronic Insomnia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-02-TL-375-017; U1111-1114-8272 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramelteon and Placebo QD (9 possible combinations total) (Experimental)
  Interventions: Drug: Ramelteon and Placebo (9 possible combinations total)

INTERVENTIONS:
Drug: Ramelteon and Placebo (9 possible combinations total) — Randomized sequence over two consecutive nights for a total of three treatment periods to include the following:
  Ramelteon 4 mg, tablets, orally over two nights
  Ramelteon 8 mg, tablets, orally over two nights
  Ramelteon placebo-matching tablets, orally over two nights
  Other Names: Ramelteon; Rozerem; TAK-375

SUMMARY:
This purpose of this study is to assess the efficacy and safety of Ramelteon, once daily (QD), in elderly subjects with chronic insomnia.

DETAILED DESCRIPTION:
Insomnia is characterized by a complaint of difficulties initiating and maintaining sleep or of nonrestorative and non-refreshing sleep. Transient insomnia affects approximately one-third to one-half of the US population, based on the results of 2 surveys of representative samples of the adult US population conducted by the Gallup Organization in which respondents were asked if they had .ever had difficulty sleeping. Based on reports of regular or frequent sleep difficulty, results from the same studies suggest that approximately one-tenth of the US population experiences chronic insomnia. The ideal treatment for insomnia would reduce the latency to onset of sleep and increase total sleep time, without a negative impact on sleep architecture and without safety concerns or next-day effects.

Ramelteon is a melatonin-1 receptor agonist under global development by Takeda Chemical Industries, Ltd., Osaka, Japan, for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

Participation in this study is anticipated to be about 2 months.

ELIGIBILITY:
Inclusion Criteria

* Male or a post-menopausal female.
* Primary insomnia as defined by the Diagnostic and Statistical Manual of Mental Disorders, Text Revision for at least 3 months and as defined by subjective sleep latency greater than or equal to 30 minutes, subjective total sleep time less than or equal to 6.5 hours per night, and daytime complaint(s) associated with disturbed sleep.
* Mean latency of greater than or equal to 20 minutes per polysomnography on two consecutive screening nights with neither night less than 15 minutes. Also, a mean of 60 minutes of wake time during the 480 minutes in bed across two nights with no night less than 45 minutes.
* Habitual bedtime is between 8:30 p.m. and 12:00 a.m.
* Body mass index between 18 and 34, inclusive.

Exclusion Criteria

* Known hypersensitivity to Ramelteon or related compounds, including melatonin.
* Previously participated in a study involving Ramelteon.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to Day 1 of single-blind study medication, whichever is longer.
* Sleep schedule changes required by employment (eg, shift worker) within three months prior to Day 1 of single-blind study medication, or has flown across greater than three time zones within seven days prior to screening.
* Participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to Day 1 of single-blind study medication.
* Ever had a history of seizures, sleep apnea, chronic obstructive pulmonary disease, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
* History of psychiatric disorder (including anxiety or depression) within the past 12 months.
* History of drug addiction or drug abuse within the past 12 months.
* History of alcohol abuse within the past 12 months.
* Had an acute clinically significant illness, as determined by the investigator, within 30 days prior to Day 1 of single-blind study medication.
* Current significant neurological (including cognitive and psychiatric disorders), hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, or metabolic disease, unless currently controlled and stable with protocol-allowed medication 30 days prior to Day 1 of single-blind study medication.
* Used tobacco products within 90 days prior to Day 1 of single-blind study medication.
* Used melatonin, or other drugs or supplements known to affect sleep/wake function, or has consumed grapefruit or grapefruit juice within 5 days (or 5 half lives, whichever is longer) prior to Day 1 of single-blind study medication.
* Used any central nervous system medication within 3 weeks (or 5 half lives of the drug, whichever is longer) prior to Day 1 of singleblind study medication. These medications must not have been used to treat psychiatric disorders.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel including anti-hepatitis A virus (only immunoglobulin M is exclusionary), anti- hepatitis B surface (except in subjects who have received hepatitis B virus vaccination), hepatitis B surface antigen, anti- hepatitis B core (only immunoglobulin M is exclusionary), or anti-hepatitis C virus.
* Positive urine drug screen including alcohol at screening and each check-in or a positive breathalyzer test at each check-in.
* Apnea hypopnea index (per hour of sleep) greater than 15 as seen on polysonography, on the first night of the polysonography screening.
* Periodic leg movement with arousal index (per hour of sleep) greater than 20 as seen on polysonography, on the first night of polysonography screening.
* Any additional condition(s) that in the Investigator.s opinion would: a) affect sleep/wake function, b) prohibit the subject from completing the study, or c) not be in the best interest of the subject to participate in the study.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Within 3 weeks prior to Day 1 of single-blind study medication and during the study:

    * anxiolytics
    * hypnotics
    * antidepressants
    * anticonvulsants
    * sedating H1 antihistamines
    * systemic steroids
    * respiratory stimulants (eg, theophylline) and decongestants
    * over-the counter and prescription stimulants
    * over-the counter and prescription diet aids
    * central nervous system active drugs (including herbal preparations with central nervous system effects)
    * narcotic analgesics
    * beta blockers
    * St. John.s wort
    * kava-kava
    * gingko biloba, any other supplements
  * Within 5 days prior to Day 1 of single-blind study medication and during the study:

    * melatonin, or other drugs or supplements known to affect sleep/wake function.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-10; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Mean latency to persistent sleep of 2-night per polysomnogram recordings, from nights 1 and 2 of each Treatment Period. | Crossover Periods 1, 2, and 3 on Nights 1 and 2 or Final Visit.

SECONDARY OUTCOMES:
Total Sleep Time. | Crossover Periods 1, 2, and 3 on Nights 1 and 2 or Final Visit.
Sleep Efficiency. | Crossover Periods 1, 2, and 3 on Nights 1 and 2 or Final Visit.
Wake Time after Sleep Onset. | Crossover Periods 1, 2, and 3 on Nights 1 and 2 or Final Visit.
Number of Awakenings after Persistent Sleep Onset. | Crossover Periods 1, 2, and 3 on Nights 1 and 2 or Final Visit.
Subjective Sleep Latency. | Crossover Periods 1, 2, and 3 on Mornings 2 and 3 or Final Visit.
Subjective Total Sleep Time. | Crossover Periods 1, 2, and 3 on Mornings 2 and 3 or Final Visit.
Subjective Wake Time after Sleep Onset. | Crossover Periods 1, 2, and 3 on Mornings 2 and 3 or Final Visit.
Subjective Number of Awakenings. | Crossover Periods 1, 2, and 3 on Mornings 2 and 3 or Final Visit.
Subjective Ease of Falling Back to Sleep after Awakening. | Crossover Periods 1, 2, and 3 on Mornings 2 and 3 or Final Visit.
Subjective Sleep Quality. | Crossover Periods 1, 2, and 3 on Mornings 2 and 3 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (18):
- United States (18):
  - Hot Springs, Arkansas
  - Irvine, California
  - Palm Springs, California
  - San Diego, California
  - Brandon, Florida
  - Miami, Florida
  - Naples, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Overland Park, Kansas
  - Crestview Hills, Kentucky
  - Troy, Michigan
  - St Louis, Missouri
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Houston, Texas

REFERENCES:
- [Result] Roth T, Seiden D, Wang-Weigand S, Zhang J. A 2-night, 3-period, crossover study of ramelteon's efficacy and safety in older adults with chronic insomnia. Curr Med Res Opin. 2007 May;23(5):1005-14. doi: 10.1185/030079907x178874. PMID 17519067
- [Result] Wang-Weigand S, McCue M, Ogrinc F, Mini L. Effects of ramelteon 8 mg on objective sleep latency in adults with chronic insomnia on nights 1 and 2: pooled analysis. Curr Med Res Opin. 2009 May;25(5):1209-13. doi: 10.1185/03007990902858527. PMID 19327100
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI